CLINICAL TRIAL: NCT00469651
Title: A Double Blind, Randomized, Controlled Phase Ib Field Trial in 12 to 24 Month Old Children in Tanzania to Evaluate the Safety and Immunogenicity of Candidate Malaria Vaccine MSP 3 Versus Hepatitis B Vaccine
Brief Title: Phase Ib Trial of MSP3 LSP in Children in Tanzania
Acronym: MSP3TN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: African Malaria Network Trust (Network)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Dr. Roma Chilengi, African Malaria Network Trust
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSP3_TN_0303; MSP3 TN_03_03
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Malaria
Keywords: Malaria; vaccine; MSP3LSP; Safety; children; Tanzania
MeSH Terms: conditions — Malaria | interventions — MSP3 protein, Plasmodium falciparum (181-276); Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 15 microgramme candidate vaccine
  Interventions: Biological: MSP3 vaccine
- 2 (Active Comparator): Hepatitis B vaccine
  Interventions: Biological: Hepatitis B vaccine
- 3 (Experimental): 30 microgramme MSP3 candidate malaria vaccine
  Interventions: Biological: MSP 3 Long Synthetic Peptide; Biological: MSP3 candidate vaccine
- 4 (Active Comparator): Hepatitis B control vaccine
  Interventions: Biological: Hepatitis B control vaccine

INTERVENTIONS:
Biological: MSP 3 Long Synthetic Peptide — Lyophilized MSP3 vaccine adjuvanted in Aluminium hydroxide
  Arms: 3
Biological: MSP3 vaccine — Lyophilized vaccine adjuvanted in Aluminium hydroxide
  Arms: 1
Biological: Hepatitis B vaccine — Hepatitis B vaccine adjuvanted in Aluminium hydroxide
  Arms: 2
Biological: MSP3 candidate vaccine — Lyophilized MSP3 adjuvanted in Aluminium hydroxide
  Arms: 3
Biological: Hepatitis B control vaccine — Hepatitis B vaccine adjuvanted in Aluminium Hydroxide
  Arms: 4

SUMMARY:
This study will evaluate the safety of candidate malaria vaccine MSP3 in children aged 12-24 months in Tanzania in a highland area with low malaria transmission.

Written informed consent will be sought from all guardians/parents of potentially participating children. Eligible children will be randomly allocated to receive either the the study vaccine (MSP3 for a total of 30 children)) or the control vaccine (hepatitis B for a total of 15 children). The vaccines will be given in 3 immunizations one month apart to all the study children and neither the clinical investigators nor the children's parents will be aware of which vaccine has been administered during the initial four months of the study. The study is designed to begin with a lower dose of the MSP3 vaccine (15µg of MSP3 for 15 children) and then followed by the higher dose(30µg MSP3 for 15 children). Following each immunization, children will be evaluated for a seven day solicited symptoms. Unsolicited symptoms will also be collected throughout the study duration.

The study will be overseen by an international safety monitoring committee who will follow safety matters closely as the trial progresses. The study will also be approved by the Tanzania National ethics Committee, The Tanzania Food and Drugs Authority, and the London school of hygiene and tropical medicine ethics committee. The study is planned to last 13 months for each participant.

DETAILED DESCRIPTION:
The study is a double blind (observer blind, participant blind), randomized, controlled, dose escalation, Age deescalation, phase Ib study. It will include two parallel groups as follows:

* Group 1: 23 subjects (15 subjects receiving MSP3-LSP vaccine 15 µg and 8 subjects receiving Hepatitis B vaccine).
* Group 2: 22 subjects (15 subjects receiving MSP3-LSP vaccine 30 µg and 7 subjects receiving Hepatitis B vaccine).

The Immunization schedule will be 0, 1, and 2 months for all cohorts and provisionally as following for each group:

* Study days 0, 28 and 56 for group 1
* Study days 14, 42, 70 for group 2 Vaccinations of groups 1 and 2 will be staggered: immunization in group 2 will start 2 weeks after group 1. This interval may be extended if deemed necessary in case of serious adverse events or other safety concerns. Randomization will be done for each group at the time of first vaccinations and only the study pharmacist will be aware of which vaccine is allocated to a particular study ID number. The pharmacist will have no other role and will be sworn to confidentiality.

The study vaccine will be administered through the subcutaneous injection into right or left deltoid (alternately). Each child will be observed for at least 60 minutes after vaccination to evaluate and treat any acute adverse events.

This will be followed by a Seven (7) day follow-up period for solicited adverse events (day of vaccination plus 6 subsequent days; twenty eight (28) day follow-up period for unsolicited adverse events (Vaccination day plus 27 subsequent days). The follow-up of serious adverse events (SAE's) for 12 months after the first dose of study vaccine (9 months after dose 3). Biological safety will be evaluated through regular physical examinations, blood sampling for routine clinical chemistry, and hematology). At the end of the follow-up period for unsolicited AEs (i.e., one month after the third dose), children will be followed by field workers at home at monthly intervals to record SAEs. There are 10 clinic visits planned, however, participants will be advised to report to the clinic any time they feel unwell.

Data collection will be through participant record files from which transcription on to conventional Case Report Forms will be done. All the date on the CRFs will be verified by the clinical Monitor. The database will be locked after study day 84 to allow for an interim analysis to review safety and immunogenicity thus collected.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-2 years old
* Healthy by medical history and physical examination
* Signed /thumb printed informed Consent by guardian/parent
* Resident in the study area village during the whole trial period

Exclusion Criteria:

* Symptoms, physical signs of disease that could interfere with the interpretation of the trial results or compromising the health of the subjects.
* Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior recruitment (for corticosteroids, this means prednisolone or equivalent 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Cannot be followed for any social, psychological or geographical reasons.
* Use of any investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose.
* Suspected or known hypersensitivity to any of the vaccine components or to previous vaccine.
* Laboratory abnormalities on screened blood samples out of range, more specifically refer to table 4.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine. An exception is the receipt of an EPI or licensed vaccine (measles, oral polio, meningococcal and combined diphtheria/pertussis/tetanus vaccines) which may be given 14 days or more before or after vaccination.
* Evidence of chronic or active Hepatitis B infection.
* Presence of chronic illness that, in the judgment of the investigator, would interfere with the study outcomes or pose a threat to the participant's health.
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of surgical splenectomy.
* Moderate or severe malnutrition at screening defined as weight for age Z-score less than 2

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2007-10; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Safety of MSP3 by assessing the reactogenicity | Solicited and unsolicited adverse events (immediate reactogenicity within 60 minutes of each vaccination; 7-day assessment, and 28 days

SECONDARY OUTCOMES:
The humoral response to vaccine antigens will be assessed by measuring by ELISA | ELISA on D0, D28, D56, D84, D168 and D365

CONTACTS AND LOCATIONS:
Overall Officials: Martha M Lemnge, MS, PhD, Study Director — National Institute For Medical Research in Tanzania; John P Lusingu, MD, PhD, Principal Investigator — National Institute for Medical Research in Tanzania
Locations (1):
- Kwashemshi village, Korogwe, Tanga, Tanzania

REFERENCES:
- [Derived] Lusingu JP, Gesase S, Msham S, Francis F, Lemnge M, Seth M, Sembuche S, Rutta A, Minja D, Segeja MD, Bosomprah S, Cousens S, Noor R, Chilengi R, Druilhe P. Satisfactory safety and immunogenicity of MSP3 malaria vaccine candidate in Tanzanian children aged 12-24 months. Malar J. 2009 Jul 17;8:163. doi: 10.1186/1475-2875-8-163. PMID 19607731